CLINICAL TRIAL: NCT06472609
Title: Prospective Quality Improvement Project for High-Risk Diabetes Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Close-out meeting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: N202105025
Record Dates: First submitted 2023-05-26; First posted 2024-06-25 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus; Latent Tuberculosis Infection; Continuous Glucose Monitoring; Quality of Life
Keywords: Diabetes Mellitus; Quality of Life; Latent Tuberculosis Infection; Continuous Glucose Monitoring
MeSH Terms: conditions — Diabetes Mellitus; Latent Tuberculosis

STUDY DESIGN:
Intervention Model Description: Diabetic patients have had poor blood glucose control in the past year, and have a record of glycated hemoglobin (HbA1C%) greater than 9%.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- interactive group (Experimental): diabetes, enhanced interactive education program through weekly phone call for 12 weeks
  Interventions: Behavioral: enhanced interactive education

INTERVENTIONS:
Behavioral: enhanced interactive education — The present study is a prospective randomized open-label study. Patients with diabetes mellitus who have HbA1c% more than 9% during the recent 1 year are enrolled. The intervention group receives, besides routine medical control of diabetes,enhanced interactive education program through weekly phone call for 12 weeks.

SUMMARY:
Diabetes is the most important comorbidity of tuberculosis patients in Taiwan, and 1/4 of tuberculosis patients also It is a diabetic patient, and the treatment of latent tuberculosis infection is currently an important policy of the Taiwan Disease Control Agency One, because babies are prone to encounter difficulties in the early stages, because of the spread of Australian patients in the community, The Department of Disease Control encourages patients with diabetes to receive screening and treatment for latent tuberculosis infection.

DETAILED DESCRIPTION:
Diabetes mellitus is the most prevalent comorbiditiy for patients with active tuberculosis in Taiwan. More than one fourth of the patients with incident tuberculosis has diabetes mellitus. The latent tuberculosis infection treatment is recommended by the Centers of Disease Control (CDC) of Taiwan to halt the transmission of tuberculosis in the community. Considering a relatively long delay in diagnosis of tuberculosis in clinical practice, eliminate the dormant tuberculosis germs a the stage of latent infection is the most cost-effective strategy to avoid tuberculosis transmission. The population with diabetes mellitus and inadequate blood sugar control are at increased risk of latent tuberculosis infection and activation and are encouraged to undergo latent tuberculosis screening and treatment. However, the anti-tuberculosis agents could have significant drug-drug interaction with the drugs used for diabetes mellitus control. The extent of its impact on blood sugar is still unclear. We aim to investigate the fluctuation of blood sugar during latent tuberculosis treatment with continuous subcutaneous sugar monitoring device to evaluate the possible associated risk of hyperglycemia or hypoglycemia to enhance treatment safety. Inadequate blood sugar control is the root for immune dysfunction and render the patients vulnerable to infectious diseases. Hence, improvement in the blood sugar control not only leads to a better immune function to avoid tuberculosis infection but also reduce the risk of progression for cardiovascular and renal disorder. The present study proposed a protocol of 12-week aggressive blood sugar control and education program using phone call to improve the blood sugar control and life quality. Furthermore, to evaluate the efficacy of anti-tuberculosis treatment for latent tuberculosis, we propose to evaluate the mycobacteria-specific antigen immune response by using the interferon-gamma releasing assay before and after anti-tuberculosis treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients had a record of glycated hemoglobin (HbA1C%) greater than 9% in the past year.

Exclusion Criteria:

* Be younger than 20 years old.
* Unconsciousness or severe dementia, unable to conduct quality of life questionnaire assessment.

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2021-07-29 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
quality improvement project | 12 weeks
  After the admitted patients were involved in the quality improvement project, the glycated blood demand in the 12 weeks was tracked as the target index for purposeful control and research, and the final value was compared.
  The quality of life of the case was evaluated by using the Diabetes-Related Distress Questionnaire (DRDQ) as an evaluation index to compare the differences before and after the intervention of the interdisciplinary care team.

SECONDARY OUTCOMES:
Immune response to tuberculosis-specific antigen. | 12 weeks
  In cases of latent tuberculosis infection, Quantiferon-Gold Plus is used to evaluate the immune response of CD8 T cell lymphocytes to tuberculosis-specific antigens before and after treatment.
Number of episodes of hyperglycemia or hypoglycemia in people with high-risk diabetes | 14 weeks
  For high-risk diabetic patients receiving treatment for latent tuberculosis infection, use a continuous blood glucose monitor to compare the incidence of adverse events such as hyperglycemia or hypoglycemia five days before and five days after medication.
quality of life measures | 12 weeks
  The quality of life of the case was evaluated by using the Diabetes-Related Distress Questionnaire (DRDQ) as an evaluation index to compare the differences before and after the intervention of the interdisciplinary care team.

CONTACTS AND LOCATIONS:
Locations (1):
- Chih-Hsin,Lee, Taipei, Taiwan, Taiwan